CLINICAL TRIAL: NCT04119297
Title: Effects of Cold Application and Heparinoid on Periorbital Edema and Ecchymosis After Craniotomy
Brief Title: Effects of Cold Application and Heparinoid on Periorbital Edema and Ecchymosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Serpil Yüksel, Assistant Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3791
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Neurological Disorder; Nursing Caries; Periorbital Edema; Ecchymosis; Cryotherapy Effect
Keywords: Cold application; Craniotomy; Heparinoid; Periorbital edema; Periorbital ecchymosis
MeSH Terms: conditions — Nervous System Diseases; Orbital Cellulitis; Ecchymosis | interventions — Isotonic Solutions

STUDY DESIGN:
Intervention Model Description: This study was conducted as a prospective, parallel, three arm (1:1:1), randomized controlled clinical trial at neurosurgical intensive care units (NICU) and neurosurgical clinics in two medical faculty hospital of a university in Istanbul, Turkey.
Who Masked: Participant, Investigator
Masking Description: The random allocation cards was developed using a computer generated random number by a biostatistician who was not associated with the study. Group allocation was concealed using individual sealed opaque envelopes. As patients were enrolled in the study, the next envelope was extracted and the patients was assigned to the groups accordingly. When the patient was transferred from the operating theatre to the NICU or clinic, the nurse in the study (NA) assigned the patient to one of the groups according to the list in the envelope. Other investigator nurse (SY), two observer nurses (DG, YT), and all patients were blinded from group assignment. Also, all patients were blinded to all measurements and, the investigator and two observers were blinded to each other's measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Routine care (Irregular cold application or gauze bandages wetted with isotonic solution or once daily heparinoid cream application) of the clinic was applied.
  Interventions: Other: Routine care
- Cold application (Experimental): Cold application was applied for three days after craniotomy.
  Interventions: Other: Cold gel pack
- Heparinoid group (Experimental): Heparinoid cream was applied for three days after craniotomy
  Interventions: Drug: Heparinoids Topical Cream

INTERVENTIONS:
Other: Routine care — * Routine care was applied to the periorbital area by clinical nurses.
  * Periorbital edema, upper and lower eyelid ecchymosis of the patients were evaluated on the 3rd and 9th hours after craniotomy, and on the 1st, 2nd and 3rd days (twice daily) using the Kara & Gokalan's Scale
  Other Names: Irregular cold application or gauze bandages wetted with isotonic solution or once daily heparinoid cream application
  Arms: Control
Other: Cold gel pack — * Cold application was applied to the periorbital area for 20 minutes per hour beginning 3rd hour following craniotomy, except from 10pm-7 am, and for three days using gel pack cooled to -14ºC.
  * Periorbital edema, upper and lower eyelid ecchymosis of the patients were evaluated on the 3rd and 9th hours after craniotomy, and on the 1st, 2nd and 3rd days (twice daily) using the Kara & Gokalan's Scale
  Other Names: Cold application
  Arms: Cold application
Drug: Heparinoids Topical Cream — * Heparinoid cream was applied to the periorbital area once at 3rd and 9th hours following craniotomy, and 4 times daily in the following 3 days.
  * Periorbital edema, upper and lower eyelid ecchymosis of the patients were evaluated on the 3rd and 9th hours after craniotomy, and on the 1st, 2nd and 3rd days (twice daily) using the Kara & Gokalan's Scale
  Other Names: local heparinoid application
  Arms: Heparinoid group

SUMMARY:
During surgery, blood leaking from damaged blood vessels spread to the periorbital area may cause periorbital edema and ecchymosis after anterior craniotomy. This study was carried out to determine the effects of the cold application and the local heparinoid on periorbital edema and ecchymosis after craniotomy.

DETAILED DESCRIPTION:
Periorbital edema and ecchymosis are common after anterior craniotomy. Periorbital edema and ecchymosis are not complications, they are natural outcomes of surgical trauma. However, periorbital edema prevents pupil examination and causes the patient to experience fear and anxiety with accompanying ecchymosis. Periorbital edema rate after anterior craniotomy was 36.8-100%, ecchymosis rate was 62.5%, and 30% of patients with edema did not have a pupil examination for the first 36 hours after craniotomy.The present study was carried out to determine the effects of the heparinoid creams and regular cold application performed using gel packs in controlling periorbital edema and ecchymosis after craniotomy.

ELIGIBILITY:
Inclusion Criteria: The eligible participants were those

* who were aged 18 years and older
* who had Glasgow Coma Scale score > 15
* who had no mental and physical problems that interfere with communication
* whose vital signs were normal
* who had no ptosis
* who volunteered to participate and signed the informed consent form

Exclusion Criteria:The participants excluded from the study;

* who had Glasgow Coma Scale score < 15
* who died during surgery
* ptosis formed after surgery
* who refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Periorbital edema | Evaluation was performed twice a day for three days after craniotomy.
  This edema defined as swelling around the eye was evaluated using the Kara & Gokalan's Scale.
Periorbital ecchymosis | Evaluation was performed twice a day for three days after craniotomy.
  This ecchymosis is produced by blood tracking into periorbital tissues, causing blue or purple discoloration of the upper and lower eyelid. Evaluation was performed with using the Kara & Gokalan's Scale.

SECONDARY OUTCOMES:
Periorbital superficial skin temperature | Skin temperature was measured every hour before and after cold application
  Change in periorbital superficial skin temperature after cold application

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Yüksel, PhD, Principal Investigator — Necmettin Erbakan University

IPD SHARING:
Plan to Share IPD: No